CLINICAL TRIAL: NCT00659438
Title: A Randomized, Double-blind Phase II Trial to Assess the Efficacy and Safety of Bicalutamide (Casodex® ) Associated to ZD6474 (Zactima™ ) or to Placebo in Patients With Castration-refractory Metastatic Prostate Cancer Without Any Clinical Symptom Related to Disease Progression
Brief Title: Efficacy and Safety of Zactima™ in Patients With Castration-refractory Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4200C00080; 2007-001891-35 (EudraCT Number)
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — vandetanib; bicalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Bicalutamide 150mg + ZD6474 300mg
  Interventions: Drug: ZD6474 (Vandetanib); Drug: Bicalutamide
- 2 (Placebo Comparator): Bicalutamide 150mg + placebo
  Interventions: Drug: Bicalutamide; Drug: Placebo

INTERVENTIONS:
Drug: ZD6474 (Vandetanib) — 300mg orally, once daily
  Other Names: Zactima
  Arms: 1
Drug: Bicalutamide — 150mg orally, once daily
  Other Names: Casodex
Drug: Placebo — orally, once daily
  Arms: 2

SUMMARY:
This randomized, double-blind phase II trial is to assess the efficacy and safety of bicalutamide (Casodex® ) associated to ZD6474 (Zactima™ ) or to placebo in patients with castration-refractory metastatic prostate cancer without any clinical symptom related to disease progression. The study is blinded, and subjects will be randomised (1:1 ratio) to either ZD6474 300 mg or placebo. The blinded design ensures robust, unbiased data collection and assessment. Placebo control is necessary to ensure a robust assessment of PSA PFS, and is acceptable in this subject population where all subjects will also received bicalutamide 150 mg o.d. Subjects will continue study treatment until they reach objective biological disease progression or unacceptable toxicity or withdrawal of consent or until end of trial (which event occurs first). The end of study is fixed 12 months after the last randomised patient's first dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males presented with a confirmed histological diagnosis of adenocarcinoma of the prostate with evidence of metastases (including bone, lymph nodes, or other site) radiologically or histologically documented and despite a serum testosterone ≤1.73 nmol/L (50 ng/dL) proving castration, evidence of biochemical progression of prostate cancer, documented by a rise in PSA .

Exclusion Criteria:

* Radiotherapy or surgery or antiandrogens (except LHRH analogue) or bilateral orchiectomy within the 30 days preceding Visit 1. Incompletely healed surgical incision.
* Concomitant anticancer therapy other than surgical castration or continuous medical castration.
* Biology restriction.
* Clinical significant cardiovascular event or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
* History of arrhythmia which is symptomatic or requires treatment (CTCAE grade 3), symptomatic despite treatment, or asymptomatic sustained ventricular tachycardia. Subjects with atrial fibrillation controlled on medication are permitted.
* Hypertension not controlled by medical therapy
* ECG /QTc prolongation
* Presence of left bundle branch block (LBBB).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2008-02; Primary Completion 2010-11 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- France (5):
  - Research Site, Bordeaux
  - Research Site, Créteil
  - Research Site, Paris
  - Research Site, Reims
  - Research Site, Villejuif

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 4th, 2008 to April 26th, 2010, 8 centers in France.
Pre-assignment Details: 110 participants screened; 95 participants were randomized to receive either bicalutamide 150 mg + vandetanib 300 mg once daily oral dose or bicalutamide 150 mg + placebo.
Groups:
- Vandetanib: Bicalutamide 150mg + Vandetanib (ZD6474) 300mg
- Placebo: Bicalutamide 150mg + placebo
Period: Overall Study
Arm/Group | Vandetanib | Placebo
Started | 47 | 48
Assessable Set : Primary Analysis | 44 | 45
Secondary Analysis Set | 47 | 48
Safety Analysis Set | 48 (One patient randomized to placebo was accounted in vandetanib group as he mistakenly received drug) | 47
Completed | 33 | 40
Not Completed | 14 | 8
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Death | 11 | 6
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib | Placebo | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.77 (7.68) | 72.23 (6.92) | 71.51 (7.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 47 | 48 | 95

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Progression Free Rate at 4 Months
Description: To assess the effect of vandetanib on biological progression free rate based on PSA level (assessable set).
  PSA progression free rate defined as the number of participants with :
  * After decline from baseline: a 25% increase above the nadir
  * No decline from baseline: a 25% increase above the baseline (min. increase of 2 ng/mL)
Time Frame: 4 months
Measure: Number; unit: Participants
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 44 | 45
Participants | 8 | 7

2. Secondary Outcome: Progression Free Survival (PFS) at 4 Months (Instead of Time to PSA Progression)
Description: Due to the difficulties to assess biological progression date when clinical progression has occurred first, and because of the non-assessment of the clinical progression after treatment discontinuation, Time to PSA progression was not evaluated. PFS was evaluated instead, whether biological or clinical progression.
Time Frame: 4 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 47 | 48
weeks | 12.2 [11.8 to 12.4] | 12.8 [12.2 to 13.6]

3. Secondary Outcome: Progression Free Survival (PFS) at 4 Months (Instead of Time to Onset of Cancer-related Symptoms)
Description: Due to the difficulties to assess biological progression date when clinical progression has occurred first, and because of the non-assessment of the clinical progression after treatment discontinuation, Time to onset of cancer-related symptoms was not evaluated. PFS was evaluated instead, whether biological or clinical progression.
Time Frame: 4 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 47 | 48
weeks | 12.2 [11.8 to 12.4] | 12.8 [12.2 to 13.6]

4. Secondary Outcome: PSA Response Rate
Description: To investigate the effect of vandetanib on the PSA response rate. PSA response rate defined by the number of participants with a PSA decrease relative to baseline of at least 50%.
  A minimum decrease of 2 ng/mL in absolute value and a confirmation on at least 2 consecutive occasions (at least 4 weeks apart) were requested.
Time Frame: 4 months
Measure: Number; unit: Participants
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 47 | 48
Participants | 3 | 5

5. Secondary Outcome: Overall Survival (OS)
Description: To investigate the effect of vandetanib on overall survival. Patients alive at the time of the statistical analysis were censored at the time they were last known to be alive. Due to censored data, median overall survival in the placebo group cannot be calculated. OS defined as the number of participants who were alive.
Time Frame: End of study (July 2011)
Measure: Number; unit: participants
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 47 | 48
participants | 32 [lower limit 24.2] | 35

6. Secondary Outcome: Progression Rate From the Radionuclide Bone Scanning
Description: To describe the effect of vandetanib on progression rate from the radionuclide bone scanning in a sub-group of patients who had a bone scan within 3 to 6 months after 1st treatment dose. Number of participants with at least 2 new lesions on the radionuclide bone scan compared to baseline assessment were counted for calculation of progression rate.
Time Frame: 4 months
Measure: Number; unit: Participants
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 10 | 13
Participants | 3 | 4

7. Secondary Outcome: Number of Circulating Tumour Cells (CTC) (in Patients Included in Ile de France Centres Only)
Description: To investigate the effect of vandetanib on CTC. Numbering of CTCs to be performed at baseline, 1 week, 1 and 2 months after randomisation. This study was proposed only to patients followed in a study centre located in Ile de France.
  Correlation between the number of CTCs and PSA response was to be estimated after 1 week, 1 and 2 months of treatment
Time Frame: 4 months
Population: This part of the study was proposed only to patients followed in one study centre located in Ile de France and finally no blood sample has been taken at this centre. So no data on CTCs, CECs were collected and no analysis was performed.
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Circulating Endothelial Cells (CEC) of Tumour Blood Cells (in Patients Included in Ile de France Centres Only)
Description: To investigate the effect of vandetanib on CEC. Numbering of CECs was to be performed at baseline, 1 week, 1 month and 2 months after randomisation.
  Correlation between the number of CECs and PSA response was to be estimated after 1 week, 1 month and 2 months of treatment.
Time Frame: 4 months
Population: as for outcome 7
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Patients With CECs, CTCs and Gene Signature Profile of CTCs
Description: To investigate the relationship between response to vandetanib, CTCs and CECs. To investigate gene signature profile of antiangiogenic response by gene micro-array analysis of CTCs.
  Gene signature profile of CTCs was aimed to be compared before and after 2 months of treatment. No blood sample has been taken for the study, and so results on CTCs, CECs of tumour vessels and gene and signature profiles of CTCs were not performed.
Time Frame: 4 months
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Safety analysis set is composed with all randomized subjects who received at least one dose of treatment. One patient mistakenly received vandetanib during 3 days while randomized to placebo. This patient was accounted in the vandetanib group in the safety population. So, safety analysis set is composed with 48 Vandetanib and 47 placebo patients.
Arm/Group | Vandetanib | Placebo
Serious Adverse Events (participants affected / at risk) | 17/48 | 4/47
Other Adverse Events (participants affected / at risk) | 47/48 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=48) | Placebo (N=47)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Death (General disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Torsade de pointes (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Stent placement (Surgical and medical procedures) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Disease progression (General disorders) | 1 | 0
Performance status decrease (General disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=48) | Placebo (N=47)
Fatigue (General disorders) | 2 | 3
Asthenia (General disorders) | 20 | 19
Diarrhoea (Gastrointestinal disorders) | 21 | 5
Constipation (Gastrointestinal disorders) | 8 | 8
Nausea (Gastrointestinal disorders) | 9 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Hot flush (Vascular disorders) | 11 | 11
Hypertension (Vascular disorders) | 14 | 5
Dizziness (Nervous system disorders) | 5 | 5
Insomnia (Psychiatric disorders) | 4 | 6
Anxiety (Psychiatric disorders) | 2 | 7
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 5 | 0
Electrocardiogram QT prolonged (Investigations) | 8 | 1
Weight decreased (Investigations) | 5 | 1
Gynaecomastia (Reproductive system and breast disorders) | 7 | 4
Chest pain (General disorders) | 0 | 3
Pain (General disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Urinary tra ct infection (Infections and infestations) | 4 | 1
Rhinitis (Infections and infestations) | 1 | 3
Headache (Nervous system disorders) | 3 | 4
Sciatica (Nervous system disorders) | 3 | 1
Depression (Psychiatric disorders) | 4 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Haematuria (Renal and urinary disorders) | 2 | 3
Pollakiuria (Renal and urinary disorders) | 2 | 3
Dysuria (Renal and urinary disorders) | 1 | 3
Cytolytic hepatitis (Hepatobiliary disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.